CLINICAL TRIAL: NCT04687332
Title: Immunoadsorption or Plasma Exchange - What is the Best Treatment Option of Steroid Refractory Neurological Autoimmune Diseases
Brief Title: IA or PE - What is the Best Treatment Option of Steroid Refractory Neurological Autoimmune Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Mainz (Other)
Responsible Party: Principal Investigator, Prof. Dr. Julia Weinmann-Menke, Head of the Department of Nephrology and Dialysis, University Medical Center Mainz
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IA vs PE
Record Dates: First submitted 2020-12-05; First posted 2020-12-29 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Neurological Autoimmune Diseases
Keywords: Plasma exchange (PE); immunoadsorption (IA); multiple sclerosis; neuromyelitis optica,; chronic inflammatory demyelinating polyneuropathy; acute inflammatory demyelinating polyradiculoneuropathy; autoimmune encephalitis
MeSH Terms: conditions — Multiple Sclerosis; Neuromyelitis Optica; Polyradiculoneuropathy, Chronic Inflammatory Demyelinating; Guillain-Barre Syndrome; Autoimmune Diseases of the Nervous System

STUDY DESIGN:
Intervention Model Description: prospective controlled monocentric observational study
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- plasma exchange (Experimental): patients were treated with plasma exchange
  Interventions: Other: Apheresis therapy by Octo Nova Technology (DIAMED, Cologne, Germany)
- immunadsorption (Experimental): patients were treated with immunadsorption
  Interventions: Other: Apheresis therapy by Octo Nova Technology (DIAMED, Cologne, Germany)

INTERVENTIONS:
Other: Apheresis therapy by Octo Nova Technology (DIAMED, Cologne, Germany) — One group was treated with IA and the single use tryptophan adsorber, the other group was treated with PE and the Plasmaflow (see above). In total, all patients receive 5 treatments.
  Other Names: IA treatment: using single-use tryptophane adsorber TR 350 in combination with the OP-0,5W plasma separator (Asahi Kasei Medical, Tokyo, Japan) and the tubing system PA-420; PE treatment: using Plasmaflow OP 0,5W (L) and the tubing system AV-120 and FS-250

SUMMARY:
In this prospective controlled monocentric observational study, we assessed safety and efficacy of therapy with IA or PE in patients with neurological autoimmune diseases. In the subgroup analysis of MS patients also the EDSS was evaluated. In addition, we investigated possible pathomechanisms, such as cytokine alterations under therapy.

DETAILED DESCRIPTION:
Plasma exchange (PE) and immunoadsorption (IA) are first- or second line treatment options in patients with neurological autoimmune disease, including multiple sclerosis, neuromyelitis optica, chronic inflammatory demyelinating polyneuropathy, acute inflammatory demyelinating polyradiculoneuropathy (Guillain-Barré-Syndrom) or autoimmune encephalitis. This prospective controlled monocentric observational study of patients treated with either tryptophan IA or PE in cases of autoimmune neurological therapy refractory disease was performed between 2016 and 2019. The main outcome parameter for efficiency was clinical improvement after completion of treatment with PE/IA. Symptoms were assessed before the first and after the last IA/PE. In total, all patients receive 5 treatments. As patients with various neurological autoimmune diseases were included in the study, the overall treatment response was categorized descriptively as improvement or no improvement of symptoms.

ELIGIBILITY:
Inclusion Criteria:

* autoimmune neurological therapy refractory disease

Exclusion Criteria:

* Intake of Angiotensin-converting-enzyme inhibitors (ACE inhibitors) because of allergic reactions by using tryptophan adsorber
* contraindication for any anticoagulation
* contraindication for treatment with citrate dextrose anticoagulation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2019-09-15 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Change in descriptive characterization of Symptoms | After 7 days. Symptoms were assessed at baseline before the first intervention (day 1) and immediately after the last intervention (day 7).]
  Patients with various neurological autoimmune diseases were included in the study, the overall treatment response was categorized descriptively as improvement or no improvement of symptoms.
Change in the "Expanded Disability Status Scale" (EDSS) | After 7 days. EDSS were assessed at baseline before the first intervention (day 1) and immediately after the last intervention (day 7).
  In the subgroup of MS patients, disability was evaluated by EDSS. The Expanded Disability Status Scale is a scale system for the systematic recording (assessment) of disability in neurological patients suffering from multiple sclerosis. The scale is used to classify the severity of disability by symptoms, ranging from 0 (no symptoms) to a maximum of grade 10 (death from MS).

SECONDARY OUTCOMES:
Change in concentration of Immunglobulins | After 7 days. Immunglobulins were measured before and after the first intervention (day 1) and immediately before after the last intervention (day 7).
  Measurement of IgE, IgM, IgG levels and IgG subclasses.
Change in concentration of human cytokines | After 7 days. Cytokines were measured before and after the first intervention (day 1) and immediately before and after the last intervention (day 7).
  Measurement of IL-12, IL-17, IL-18, CSF-1, IL-34, IL-6, TNF-alpha and IL-28.

CONTACTS AND LOCATIONS:
Locations (1):
- UNIVERSITÄTSMEDIZIN der Johannes Gutenberg-Universität Mainz I. Medizinische Klinik und Poliklinik, Mainz, Rhineland-Palatinate, Germany